CLINICAL TRIAL: NCT03955341
Title: Clinical Evaluation and Microbiological Assessment of Diode Laser and Chemical Disinfection in Comparison to Selective Caries Removal in Management of Patients With Deep Carious Lesions: A Clinical Pilot Study
Brief Title: Clinical Evaluation and Microbiological Assessment of Diode Laser and Chemical Disinfection in Comparison to Selective Caries Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIU-IRB -1819-074
Record Dates: First submitted 2019-05-08; First posted 2019-05-20 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2020-09

CONDITIONS: Patients With Deep Carious Lesions
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: evaluate the clinical outcome (in terms of maintaining pulp vitality, assessed by cold pulp testing, absence of spontaneous pain, sensitivity to percussion, inspection for sinus or fistula or swelling, and radiographically using cone beam computed tomography) and the antimicrobial effect of Diode laser and chemical disinfection in comparison to conventional selective caries removal without disinfection in management of deep carious lesions in permanent posterior teeth.
Who Masked: Outcomes Assessor
Masking Description: Single blinded as Outcome assessors will be blinded. Both, the participants and principal investigator cannot be blinded owing to the use of two obviously different methods, laser and chemical disinfection, or no disinfection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional selective caries removal without disinfection (No Intervention): After collecting the first sample of dentin, the cavity will be restored
- Diode laser disinfection (Other): After collecting the first sample of dentin as described above, the cavity will be disinfected using Diode laser (EPIC™, BIOLASE) with 940 nm and an output power of 0.5 watt (24). A 400 µm noninitiated tip will be used for cavity irradiation, in a noncontact mode (2mm distance), 5 sec/mm2 in sweeping motion. A 2nd dentinal sample will be collected after diode laser disinfection.
  Interventions: Device: Diode laser disinfection
- Chemical disinfection using 2% Chlorhexidine (Other): After collecting the first sample of dentin, the cavity will be disinfected using 2% Chlorhexidine (Consepsis®, Ultradent) for 20 seconds (32). Then a 2nd dentinal sample will be collected after chemical disinfection.
  Interventions: Other: Chemical disinfection using 2% Chlorhexidine

INTERVENTIONS:
Device: Diode laser disinfection — After collecting the first sample of dentin as described above, the cavity will be disinfected using Diode laser (EPIC™, BIOLASE) with 940 nm and an output power of 0.5 watt (24). A 400 µm noninitiated tip will be used for cavity irradiation, in a noncontact mode (2mm distance), 5 sec/mm2 in sweeping motion. A 2nd dentinal sample will be collected after diode laser disinfection.
  Arms: Diode laser disinfection
Other: Chemical disinfection using 2% Chlorhexidine — After collecting the first sample of dentin, the cavity will be disinfected using 2% Chlorhexidine (Consepsis®, Ultradent) for 20 seconds (32). Then a 2nd dentinal sample will be collected after chemical disinfection.
  Arms: Chemical disinfection using 2% Chlorhexidine

SUMMARY:
Objectives: To evaluate the clinical and antimicrobial effect of Diode laser and chemical disinfection in comparison to selective caries removal in management of deep carious lesions.

Methods: This study will be carried on 30 patients with an age range of 18 -50 years. The patients will be selected from the outpatient clinics in Faculty of Oral and Dental Medicine, Misr International University. All patients will be randomly divided into 3 equal groups; Control group, Diode laser application with an output power of 0.5 watt group, and Chemical disinfection group. Preoperative clinical assessment and radiographs will be performed before intervention and then the patients will receive their treatment and final restorations. Follow-up with clinical assessments will be performed after 3 and 6 months. Cone beam computed tomography will be performed at the day of intervention and after 6 months. Clinical, Microbiological and Radiographic data will be collected, tabulated and statistically analyzed to compare between the success rates of diode laser, chemical disinfection and conventional selective caries removal.

DETAILED DESCRIPTION:
IV. Description of research question (PICO Question or its modifications)

PICO Question:

In management of patients with deep carious lesions in permanent posterior teeth, will the use of Diode laser with an output power of 0.5 watt or chemical disinfection using 2% Chlorhexidine affect the pulp vitality compared to conventional selective caries removal without disinfection?

Patient/Problem Patients with deep carious lesions in permanent posterior teeth

Intervention 1-Diode laser disinfection and 2- Chemical disinfection using 2% Chlorhexidine

Comparator Selective conventional caries removal without disinfection

Outcome Pulp vitality

Setting(Where will the study be performed) Dental Clinics Complex, Misr International University, and Research Unit Microbiology Lab Time (follow-up periods) 3 months and 6 months

V. Aim of the Study, Research Objectives and Clinical Relevance Aim: the aim of this study is to evaluate the clinical outcome (in terms of maintaining pulp vitality, assessed by cold pulp testing, absence of spontaneous pain, sensitivity to percussion, inspection for sinus or fistula or swelling, and radiographically using cone beam computed tomography) and the antimicrobial effect of Diode laser and chemical disinfection in comparison to conventional selective caries removal without disinfection in management of deep carious lesions in permanent posterior teeth.

Research null hypothesis:

There's no difference between the effect of Diode laser or chemical disinfection in maintaining pulp vitality compared to selective caries removal in management of deep carious lesions in permanent teeth.

* Objectives of the study:

  1. To compare the effect of diode laser versus conventional selective caries removal in maintaining pulp vitality expressed as a binary variable (success/failure), and assessed by cold pulp testing, absence of spontaneous pain, sensitivity to percussion, inspection for sinus or fistula or swelling.
  2. To compare the effect of chemical disinfection versus conventional selective caries removal in maintaining pulp vitality expressed as a binary variable (success/failure), and assessed by cold pulp testing, absence of spontaneous pain, sensitivity to percussion, inspection for sinus or fistula or swelling.
  3. To evaluate dentin thickness and density as measured by cone beam computed tomography (CBCT) using Hounsfield unit, after placement of the restorative material and at 6 months follow-up.
  4. To evaluate microbiological count in all study groups as measured by colony counter using colony-forming unit as the measuring unit.
  5. • Clinical relevance: Diode laser could yield to better clinical outcomes in management of deep carious lesions, minimizing the need for root canal treatment. This would decrease the number of treatment visits, saving time, effort, and money for both the patient and the dentist.

     Also, this leads to price reduction by decreasing the number of procedures and visits needed.

     VI. Study Design Pilot clinical study

     VII. Materials/ Participants (Subjects) and Methods
* Study setting: Study is to be conducted in Dental Clinics Complex (MIU Dental Laser Center) in Misr International University, Egypt.

Patients are to be selected from the outpatient dental clinics complex, Misr International University.

The microbiological testing will be performed at the Bacteriology lab, Research unit, MIU Sample type:

Purposive sample

Method of randomization:

Computer generated randomization for sequence will be held at the 1st visit. Randomization will be performed through computed software (www.randomizer.org).

The number corresponding to each treatment procedure will be recorded on cards kept inside sequentially numbered, opaque, sealed envelopes.

• Sample size calculation: Due to lack of sufficient literature and this is the first study to our knowledge evaluating the primary outcome (pulp vitality), after using diode laser disinfection. Thus, this pilot study will be carried out on 30 patients. So, each group will include 10 patients. Sample size power will be calculated based on the results of this pilot study using G*Power Version 3.1.9.2 to continue full sample size.

1. Statistical Analysis

1. Clinical, microbiological and radiographic data will be collected, tabulated and statistically analyzed to compare between the success rates of diode laser, chemical disinfection, and selective caries removal, using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation, while qualitative data will be described as number and percentage.
2. Comparisons between the study groups will be performed using suitable parametric and non-parametric tests of significance depending on the distribution of the collected data.

2. Intervention (methods, blinding)

I-) Operative procedures:

The procedures involve performing conservative caries management for one tooth per patient, using either Diode laser or 2% Chlorhexidine (chemical disinfectant) or no disinfection (24,32). Patients will be randomly allocated into one of the three study groups using computed software (www.randomization.com); group 1: Diode laser disinfection with an output power of 0.5 watt, group 2: Chemical disinfection using 2% Chlorhexidine, and group 3: conventional selective caries removal without disinfection (control group). The same final restorative materials will be used in all groups, so that the outcome would only reflect the effect of the technique of disinfection versus no disinfection. Each patient will be assessed for eligibility, the procedures will be explained to him/her and if they agree to participate, they sign the informed consent form.

* The principal investigator will perform the procedures for all patients.
* Preoperative clinical assessment and periapical radiographs will be performed before starting the procedures.
* Local anesthesia will be administered and the tooth will be isolated with a rubber dam.
* Access to the lesion will be gained with a sterile high-speed bur or diamond burs, to establish the outline form.
* Caries will be completely removed from the surrounding cavity walls.
* Superficial necrotic carious fragments will be removed from the floor using a sharp sterile excavator, while soft dentin will be left on the floor to avoid pulpal exposure.

I-Dentinal sample collection:

- Samples will be collected from each patient from the base of the infected cavity using sterile using sterile spoon excavator. Sample will be transferred to sterile Eppendorf tubes containing 0.5 ml of phosphate buffer saline solution with aseptic precautions.

Group 1) (Intervention Diode laser disinfection with an output power of 0.5 watt group):

After collecting the first sample of dentin as described above, the cavity will be disinfected using Diode laser (EPIC™, BIOLASE) with 940 nm and an output power of 0.5 watt (24). A 400 µm noninitiated tip will be used for cavity irradiation, in a noncontact mode (2mm distance), 5 sec/mm2 in sweeping motion. A 2nd dentinal sample will be collected after diode laser disinfection.

Group 2) (Intervention chemical disinfection group):

After collecting the first sample of dentin, the cavity will be disinfected using 2% Chlorhexidine (Consepsis®, Ultradent) for 20 seconds (32). Then a 2nd dentinal sample will be collected after chemical disinfection.

Group 3) Comparator (Control group):

After collecting the first sample of dentin, the cavity will be restored.

* For all groups, the cavity will be filled with glass ionomer material as a base material and then will be restored with resin composite restoration.
* Patients will receive postoperative instructions and oral hygiene guidelines that should be followed during the follow-up period.
* Patients will be recalled for follow up visit after three and six months to follow-up the pulp vitality and restoration condition.
* Outcome assessment will be performed by the outcome investigators according to the evaluation chart.

II) Observations:

1. Clinical Evaluation:

   • Follow-up with clinical assessments will be performed after 3 and 6 months (T3 and T6).

   Upon completing the intervention, the patient will be recalled after 3 and 6 months to assess outcome. To assess the primary outcome (pulp vitality), previous studies have used a binary variable (success/failure) indicating whether the restored tooth maintained its vitality at the outcome investigation time(28). Success required positive results in all four tests mentioned below. In our study clinical success will be assessed using binary variables in addition to visual analogue scale by:

   1.1. Cold pulp testing: An ice-rod will be used for this test. Results should be positive or negative.

   1.2. Absence of spontaneous pain: Post-operative pain will be assessed using the visual Analogue Scale Score (VAS), which is a measurement method for subjective characteristics of pain. Respondents specify their level of agreement to a statement by indicating a position along a 10 cm line between two end-points, with the term "no sensitivity" at one end and "intolerable sensitivity" at the other end. A score from (0 to 10 is given).

   1.3. Sensitivity to percussion: (positive/negative). 1.4. Inspection for Sinus/fistula/swelling: using visual inspection (positive/negative).
2. Cone Beam Computed Tomography (CBT): CBT will be used to indicate the presence or absence of periapical radiolucencies (positive/negative), as well as evaluating the thickness and relative density of the remaining dentin below the final restoration. Using the smallest field of view available (5 cm x 5 cm).

   * Preoperative clinical assessment and radiographs will be performed before intervention and then the patients will receive their treatment and final restorations (T0).
   * Cone beam computed tomography will be performed at T0 and T6.
3. Microbiological Assessment:

The collected dentinal samples will be cultured on two types of selective media; Mitis salivurias agar will be used as a selective medium for Streptococcus mutans and Rogosa agar medium for Lactobacilli(1).

Total Viable Count Determination:

1. Preparation of serial dilutions: Six of tenfold serial dilution (from 10-1 to 10-6 ) will be prepared as working solutions as follows: i. 900 µl of sterile PBS or sterile Saline + 100 µl of the collected sample to prepare 10-1 dilution (D1) ii. After mixing the content of the D1, transfer 100 µl to the second tube containing 900 µl of sterile PBS or sterile Saline to prepare 10-2 dilution (D2).

   iii. Continue like this until preparing 10-6 dilution (D6). Tube Dilution Factor Dilution 1 10-1 1/10 2 10-2 1/100 3 10-3 1/1,000 4 10-4 1/10,000 5 10-5 1/100,000 6 10-6 1/1,000,000
2. Disperse 100 µl of diluted microbial solution on the surface of the plate for each selective media mentioned previously.
3. All the Rogosa agar plates will be cultured under anaerobic conditions (anaerobic gas mixture, 80% N2, 10% CO2, 10% H2) while Mitis salivurias agar plates will be cultured under aerobic conditions. Both media will be incubated at 37 °C from 24 to 48 hrs.
4. Counting bacterial colonies: Select plates that appear to have between 30 - 300 colonies in and on the agar as this gives the best statistical representation of the number of bacteria. The total number of the viable bacteria equals the number of counted colonies divided by the dilution, for example: number of colonies÷ 1/1000 (10-3) = number of colonies× 1000 • Blinding: Single blinded as Outcome assessors will be blinded. Both, the participants and principal investigator cannot be blinded owing to the use of two obviously different methods, laser and chemical disinfection, or no disinfection.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Between 18-50 years old.
  * Gender: both male and female.
  * Patients consulting in the MIU outpatient clinic.
  * Able to tolerate necessary restorative procedures (anesthesia, cavity preparation, and restorative material placement).
  * Provide informed consent.
  * Accepts the 6 months follow-up period.

Tooth related criteria:

* Permanent posterior teeth with primary deep carious lesions involving 2/3 of the entire dentin thickness with no continuity between the carious cavity and the pulp chamber, as assessed by conventional periapical radiographs.
* Teeth are vital according to pulp-sensitivity tests.

Exclusion Criteria:

* Patient-related criteria:

  1. Medically compromised patients.
  2. Pregnant women.
  3. Allergy to any of the restorative materials, including anesthetics.
  4. Uncooperative patients.

Tooth-related criteria:

1. Deciduous teeth.
2. Teeth with previous restorations.
3. Spontaneous pain or prolonged pain (more than 2 minutes) after sensitivity tests (cold and electrical tests).
4. Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion before signing the consent form.
5. Teeth presenting external or internal resorption, with adverse pulpal reactions.
6. Teeth with cervical caries.
7. Teeth showing signs of periodontitis following AAP 2017 criteria.

3. Justification of Exclusions:

Patient-related:

1. Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.
2. Pregnant women; as radiographs cannot be taken for them.
3. Allergy to any of the restorative materials, including anesthetics.
4. Uncooperative patients will not abide by the instructions or attend the appointments.

Tooth-related:

1. Deciduous teeth; as the study is targeting only permanent teeth.
2. Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
3. Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests), which would indicate irreversible pulpal damage.
4. Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion, which would indicate pulp necrosis before signing the consent form.
5. Teeth presenting external or internal resorption, with adverse pulpal reactions, which may affect the outcome of the study.
6. Teeth with cervical caries; which can't be evaluated on periapical radiographs.
7. Teeth showing signs of periodontitis following AAP 2017 criteria, which may affect the outcome of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Maintaining pulp vitality | ''through study completion, an average of 6 months"
  measuring device
  1.Cold pulp test Binary (Success/failure) If it is +ve considered success. If it is -ve, considered failure

SECONDARY OUTCOMES:
Remaining dentin density | "6 months"
  Cone Beam Computed Tomography
Reducing microbiological count | "up to 1 week"
  Colony counter

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The original data will be entered in secured database and data will be printed and saved in a secure locker to be shared with supervisors for reviewing and then to the biostatistian for statistical analysis.